CLINICAL TRIAL: NCT07100509
Title: Major Vascular Injuries in Elective Thoracic Surgery: A Single-Center 10-Year Experience
Brief Title: Major Vascular Injuries in Elective Thoracic Surgery: A 10-Year Single-Center Experience
Status: Completed | Type: Observational
Sponsor: Caner İşevi, MD (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, MD, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/ 481
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Thoracic Surgery; Vascular Injury; Intraoperative Complications
Keywords: Elective Thoracic Surgery; Intraoperative Bleeding; Cardiovascular Surgery; Vascular Injury
MeSH Terms: conditions — Vascular System Injuries; Intraoperative Complications; Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Intraoperative Vascular Injury: This cohort includes patients who experienced major intraoperative vascular injuries during elective thoracic surgeries between January 2015 and December 2024. All patients underwent surgical repair of the injured vessel, such as primary suturing, graft interposition, or ligation. No randomization or intervention assignment was performed. Data were collected retrospectively from medical records to evaluate patient characteristics, surgical details, transfusion requirements, preoperative imaging findings, complication rates, and clinical outcomes. No biospecimens were collected or retained.
  Interventions: Other: Major Vascular Injury During Elective Thoracic Surgery

INTERVENTIONS:
Other: Major Vascular Injury During Elective Thoracic Surgery — This exposure refers to patients who experienced major vascular injuries during elective thoracic surgery. Injuries involved central vessels such as the subclavian artery, brachiocephalic vein, superior vena cava, and innominate vein. No experimental intervention was applied. The study retrospectively evaluated the surgical management, transfusion requirements, preoperative planning, and clinical outcomes associated with these intraoperative events.

SUMMARY:
This study retrospectively examines major vascular injuries that occurred during elective thoracic surgeries over a 10-year period at a single tertiary care center. Although these injuries are rare, they can lead to life-threatening complications. The study aims to determine how often these injuries happen, what causes them, and how they are managed during surgery. It also evaluates the role of preoperative imaging and planning, including cardiovascular surgery team involvement, in preventing or managing these events. The findings are intended to help improve surgical safety and guide future preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective thoracic surgery between January 2015 and December 2024
* Development of a major intraoperative vascular injury during surgery
* Injury involving central vessels such as the subclavian artery or vein, brachiocephalic vein, innominate artery or vein, superior vena cava (SVC), or thoracic aorta
* Availability of complete operative and postoperative medical records
* Underwent surgical repair of the vascular injury (e.g., grafting, primary repair, ligation)

Exclusion Criteria:

* Patients undergoing emergency thoracic surgery
* Injuries limited to pulmonary artery or its branches
* Minor bleeding from peripheral vessels that did not require major intervention
* Postoperative vascular complications (e.g., delayed hemorrhage, pseudoaneurysm)
* Missing or incomplete operative records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes adult patients who underwent elective thoracic surgical procedures between January 2015 and December 2024 at a single tertiary care academic center. The study population is limited to patients who experienced major intraoperative vascular injuries involving central thoracic vessels such as the subclavian artery or vein, brachiocephalic vein, innominate artery or vein, superior vena cava (SVC), or thoracic aorta. All included patients required immediate surgical intervention for bleeding control. The study is retrospective and descriptive in nature.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Intraoperative Vascular Injuries During Elective Thoracic Surgeries | During Surgery (Intraoperative Period)
  The primary outcome is the incidence rate of major vascular injuries identified during elective thoracic surgeries performed between January 2015 and December 2024. Major vascular injury is defined as intraoperative bleeding from central vessels such as the subclavian artery or vein, brachiocephalic vein, innominate artery or vein, superior vena cava (SVC), or thoracic aorta, requiring immediate surgical intervention (e.g., primary repair, grafting, or ligation).

IPD SHARING:
Plan to Share IPD: Yes